CLINICAL TRIAL: NCT04419974
Title: Biomarkers and Genetic Modifiers in a Study of Pre-ataxic and Ataxic SCA3/MJD Carriers (BIGPRO Study) - Astrocytes
Brief Title: Astrocytic Markers and the Pre-ataxic Period of SCA3/MJD - BIGPRO Study Astrocytes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Other Study IDs: 20170014
Record Dates: First submitted 2020-04-07; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Spinocerebellar Ataxia Type 3; Machado-Joseph Disease; SCA3; MJD
Keywords: SCA3/MJD; SCA3; MJD; natural history; cytokines; astrocytes; quality of life
MeSH Terms: conditions — Machado-Joseph Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ataxic carriers: Subjects with a CAG repeat expansion on ATXN3 and Scale for Assessment and Rating of Ataxia (SARA) of 3 points or more.
  Interventions: Diagnostic Test: Clinical Scales - Baseline; Diagnostic Test: Blood Draw - Baseline; Diagnostic Test: Quality of Life Assessment - Baseline; Diagnostic Test: Clinical Scales - Follow-up 12 months; Diagnostic Test: Blood Draw - Follow-up 12 months; Diagnostic Test: Quality of Life Assessment - Follow-up 12 months; Diagnostic Test: Clinical Scales - Follow-up 24 months; Diagnostic Test: Blood Draw - Follow-up 24 months; Diagnostic Test: Quality of Life Assessment - Follow-up 24 months
- Pre-ataxic carriers: Subjects with a CAG repeat expansion on ATXN3 and Scale for Assessment and Rating of Ataxia (SARA) of less than 3 points.
  Interventions: Diagnostic Test: Molecular Diagnosis; Diagnostic Test: Clinical Scales - Baseline; Diagnostic Test: Blood Draw - Baseline; Diagnostic Test: Quality of Life Assessment - Baseline; Diagnostic Test: Clinical Scales - Follow-up 12 months; Diagnostic Test: Blood Draw - Follow-up 12 months; Diagnostic Test: Quality of Life Assessment - Follow-up 12 months; Diagnostic Test: Clinical Scales - Follow-up 24 months; Diagnostic Test: Blood Draw - Follow-up 24 months; Diagnostic Test: Quality of Life Assessment - Follow-up 24 months
- Related controls: Subjects without a CAG repeat expansion on ATXN3, but with a first degree relative affected by the disease.
  Interventions: Diagnostic Test: Molecular Diagnosis; Diagnostic Test: Clinical Scales - Baseline; Diagnostic Test: Blood Draw - Baseline; Diagnostic Test: Quality of Life Assessment - Baseline; Diagnostic Test: Clinical Scales - Follow-up 12 months; Diagnostic Test: Blood Draw - Follow-up 12 months; Diagnostic Test: Quality of Life Assessment - Follow-up 12 months; Diagnostic Test: Clinical Scales - Follow-up 24 months; Diagnostic Test: Blood Draw - Follow-up 24 months; Diagnostic Test: Quality of Life Assessment - Follow-up 24 months

INTERVENTIONS:
Diagnostic Test: Molecular Diagnosis — Double-blind molecular diagnosis for the SCA3/MJD mutation.
  Groups: Pre-ataxic carriers; Related controls
Diagnostic Test: Clinical Scales - Baseline — SARA, NESSCA, ICARS, INAS, SCAFI, CCFS will be applied on baseline.
Diagnostic Test: Blood Draw - Baseline — Blood collection on baseline for evaluation of
  * Candidate genes expression
  * Serum proteins
  * Lymphocytic proteins
Diagnostic Test: Quality of Life Assessment - Baseline — Participants fill out 2 self-reported quality of life questionnaires.
Diagnostic Test: Clinical Scales - Follow-up 12 months — SARA, NESSCA, ICARS, INAS, SCAFI, CCFS will be applied 12 months after baseline for prospective evaluation.
Diagnostic Test: Blood Draw - Follow-up 12 months — Blood collection 12 months after baseline for prospective evaluation of
  * Candidate genes expression
  * Serum proteins
  * Lymphocytic proteins
Diagnostic Test: Quality of Life Assessment - Follow-up 12 months — Participants fill out 2 self-reported quality of life questionnaires for prospective evaluation.
Diagnostic Test: Clinical Scales - Follow-up 24 months — SARA, NESSCA, ICARS, INAS, SCAFI, CCFS will be applied 24 months after baseline for prospective evaluation.
Diagnostic Test: Blood Draw - Follow-up 24 months — Blood collection 24 months after baseline for prospective evaluation of
  * Candidate genes expression
  * Serum proteins
  * Lymphocytic proteins
Diagnostic Test: Quality of Life Assessment - Follow-up 24 months — Participants fill out 2 self-reported quality of life questionnaires for prospective evaluation.

SUMMARY:
The study will consist of a prospective observation of subjects in a natural history design. The investigators will monitor changes of clinical scales, quality of life, messenger ribonucleic acid (mRNA) of candidate genes (CCL11, TNFSF14, FCGR3B, CLC, and SLA) (and their peptide products, when possible), and eotaxin and S100B serum levels, in order to determine which of them is (are) the most sensitive. Participants will be stratified in three groups: ataxic carriers, pre-ataxic carriers and non-carriers (controls).

DETAILED DESCRIPTION:
Spinocerebellar ataxia type 3, or Machado-Joseph disease (SCA3/MJD), is an autosomal dominant neurodegenerative disorder caused by a CAG expansion at ATXN3. The gene product is a 42kDa protein called ataxin-3, widely expressed in neurons and peripheral tissues. Physiological roles of ataxin-3 include, at least, ubiquitination and regulation of misfolded proteins, cytoskeletal organization and focal adhesions development, and transcriptional regulation, most often as a transcriptional corepressor. One purpose of the present study is to detect a possible association between altered transcription patterns of candidate genes and disease progression. On the other hand, previous evidences suggest that the disease process linked to polyQ aggregation in neuronal cell ("cell-autonomous process") might be worsened by what happens outside the neuronal cell ("non-cell-autonomous process"). Initial evidences lead to the role of astrocytes. This is a major depart from the traditional understanding of polyglutamine diseases, and comprises the main focus of the present study.

The main hypothesis of this study is that the SCA3/MJD clinical features may be in part associated to astrocytic processes. In order to test it, peripheral level of LIGHT protein (encoded by TNFSF14) and eotaxin (encoded by CCL11) - both expressed in astrocytes -, and of S100B (a myelin damage marker), will be measured. The investigators speculate if they can be biomarkers of disease progression and of pathological process, even before symptoms onset. In case this is positive, their responsiveness to change will be tested to check if it is better than those of clinical scales.

The second aim is to test if disease progression can be associated with changes in the transcriptional pattern of candidate genes FCGR3B, CLC and SLA.

"BIGPRO study - Astrocytes" intends to identify variations in these candidates and validate them as SCA3/MJD biomarkers. The study will consist of a prospective observation of subjects in a natural history design. Changes in clinical scales, quality of life, messenger ribonucleic acid (mRNA) of candidate genes (CCL11, TNFSF14, FCGR3B, CLC, and SLA) (and their peptide products, when possible), and eotaxin and S100B serum levels will be monitored in order to determine which of them is (are) the most sensitive. Participants will be stratified in three groups: ataxic carriers, pre-ataxic carriers and non-carriers (controls). For each asymptomatic carrier, the time until start of disease will be estimated according to the individual CAG expanded sequence (CAGexp) and subject's age. Clinical scales Scale for the Assessment and Rating of Ataxia (SARA), Neurological Examination Scale for SCA (NESSCA), International Co-operative Rating Scale (ICARS), Inventory of Non-ataxia Symptoms (INAS), SCA Functional Index (SCAFI), Composite Cerebellar Functional Severity Score (CCFS) and Quality of Life measurements (EQ-5D and SF-36), will be applied at baseline, at 12 months and at 24 months, in all subjects (all three groups). Eotaxin, TNFSF14, S100B and mRNAs, will be measured in the same moments. Progression rates of all these variables will be estimated through mixed-models, including, as covariates, age, group and their interactions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with molecular diagnosis of SCA3/MJD
* Individuals at 50% risk of inheriting SCA3/MJD mutation without any clinical manifestation

Exclusion Criteria:

* Refusal to sign informed consent
* Other diagnosed neurological conditions;
* Diabetes Mellitus;
* Chronic allergy (asthma, eczema, urticaria)
* Eosinophilia on baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with molecular diagnosis of SCA3/MJD will be recruited from the Medical Genetics Service database of Hospital de Clínicas de Porto Alegre, Brazil, by telephone calls or by invitation in the outpatient clinic. First degree relatives of these subjects at 50% risk of carrying the mutation will also be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2017-03-18 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change in serum concentrations of Eotaxin | 24 months
  pg/ml
Change in serum concentrations of S100B | 24 months
  μg/l
Change in expression of TNFSF14 | 24 months
  Fold change (FC)
Change in expression of CCL11 | 24 months
  Fold change (FC)
Change in EQ-5D-3L (EuroQoL 5 Domains evaluated in 3 levels) | 24 months
  Quality of life scale evaluating 5 domains and a visual analog scale. Domain scores increase with worsening in quality of life. In the visual analog scale, worse scores mean decrease in quality of life.
Change in SF-36 (Short-form 36) | 24 months
  Quality of life scale evaluating 8 domains through 36 questions. Domain scores decrease with worsening in quality of life.

SECONDARY OUTCOMES:
Change in expression of FCGR3B | 24 months
  Fold change (FC)
Change in expression of CLC | 24 months
  Fold change (FC)
Change in expression of SLA | 24 months
  Fold change (FC)

CONTACTS AND LOCATIONS:
Overall Officials: Laura B. Jardim, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be done via direct contact with the Principal Investigator in order to preserve individual participants identities
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will become available after final statistical analysis and data publishing via direct contact with principal investigator
Access Criteria: Investigators and researchers of the area

REFERENCES:
- See also: Official project website — https://bigpro.webnode.com/